CLINICAL TRIAL: NCT06615999
Title: Treatment Reality of Tension Band Wiring and Locked Plate Fixation of the Olecranon - Analysis of Complications, Risk Profiles and Trends
Brief Title: Treatment Reality of Tension Band Wiring and Locked Plate Fixation of the Olecranon
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Universität Münster (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. J. Christoph Katthagen, Senior Consultant, University Hospital Muenster
Other Study IDs: Olecranon TBW vs. LPF
Record Dates: First submitted 2024-09-17; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Olecranon Fracture
Keywords: Olecranon fracture; surgical treatment; locked plate fixation; tension band wiring
MeSH Terms: conditions — Olecranon Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Locking Plate fixation for simple fractured OFs (sLPF): Patients allocated to this treatment group received a locking plate fixation after the first coded diagnosis of simple fractured OF.
  Interventions: Procedure: Simple fracture locked plate fixation
- Locking Plate fixation for multi-fragmented OFs (LPF): Patients allocated to this treatment group received a locking plate fixation after after the first coded diagnosis of multi-fragmented OF.
  Interventions: Procedure: Multi-fragmented locked plate fixation
- Tension band wiring for simple fractured OFs (sTBW): Patients allocated to this treatment group received a tension band wiring fixation after the first coded diagnosis of simple fractured OF.
  Interventions: Procedure: Simple fracture Tension band wiring
- Tension band wiring for multi-fragmented OFs (TBW): Patients allocated to this treatment group received a tension band wiring fixation after the first coded diagnosis of multi-fragmented OF.
  Interventions: Procedure: Multi-fragmented tension band wiring

INTERVENTIONS:
Procedure: Simple fracture Tension band wiring — OPS 5-793.27
  Groups: Tension band wiring for simple fractured OFs (sTBW)
Procedure: Simple fracture locked plate fixation — OPS 5-793.k7
  Groups: Locking Plate fixation for simple fractured OFs (sLPF)
Procedure: Multi-fragmented tension band wiring — OPS 5-794.17
  Groups: Tension band wiring for multi-fragmented OFs (TBW)
Procedure: Multi-fragmented locked plate fixation — OPS 5-794.k7
  Groups: Locking Plate fixation for multi-fragmented OFs (LPF)

SUMMARY:
The incidence of the olecranon fracture (OF) in adults is around 12 per 100,000 inhabitants per year.1 The anatomical shape of the proximal ulna is largely responsible for the stabilization of the humeroulnar joint and reconstruction is therefore obligatory, but often challenging. Surgical treatment of the olecranon fracture is performed using tension band wiring (TBW) or locking plate fixation (LPF) osteosynthesis. It is not yet clear, which procedure is superior for a specific patient. In future, an individualized and objectified assessment of expected general and fracture-specific complications should enable the treatment to be individually adapted to the patient's risk profile. This shall prevent complications, unnecessary treatments, and treatment costs. In the project presented here, the reality of care for surgically treated patients with olecranon fractures will be analyzed using routine data collected by the BARMER health insurance fund.

The aim of the study is to analyze differences in the outcome of patients with an olecranon fracture treated with TBW compared to LPF and to identify independent risk factors for unfavorable course.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient coded diagnosis of olecranon fracture (ICD S52.01)

Exclusion Criteria:

* Incomplete basic information
* Incomplete insurance status within two years before index
* Previous treatment of olecranon fracture
* Unclear treatment of olecranon fracture
* Age < 18 years
* Coded polytrauma
* Bone tumors/ bone metastasis
* Both sides injured or missing information of surgery side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with an age of 18 years and older with an inpatient treated OF (ICD S52.01) treated with LPF or TBW between 01/2011 and 09/2023 will be included to the evaluations. Patients were grouped by age (i.e. 18-44 years, 45 - 69 years, ≥ 70 years). Younger patients (<70 years) and older patients (≥ 70 years) will be analyzed in separate studies.
Sampling Method: Non-Probability Sample
Enrollment: 15705 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Revision | up to 5 years
  Time from surgery to revision defined above.
Implant removal (only) | up to 5 years
  * Time from surgery to implant removal
  * Within first 3 months after surgery, an implant removal will also considered as a surgical complication
  * No SC is allowed to occur within 3 months and on the same day
Surgical complications (surgical complications) | up to 5 years
  Time from surgery of olecranon fracture to surgical complications, with death being considered as a competing risk event.
In-hospital surgical complication rate (IH-SC) | through hospital stay, an average of 10 days
  surgical complication after surgery during index hospitalization (yes/no)
In-hospital implant-associated complications (IH-IAC) | through hospital stay, an average of 10 days
  In-hospital implant-associated complications after surgery during index hospitalization
In-hospital non-implant associated complications (IH-non-IAC) | through hospital stay, an average of 10 days
  Non-in-hospital implant-associated complications after surgery during index hospitalizationi

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years
  * Time from surgery to death of any cause.
  * Death will be determined using the coded death as the reason for withdrawal in the BARMER database. In addition, all inpatient cases will be reviewed during follow-up, to determine whether death was reported as the reason for discharge.
30-day mortality | 30 days
  * Death from any cause within first day after surgery (yes/no)
  * All patients with shorter follow-up time are excluded
Major adverse events (MAE) | up to 5 years
  Time from surgery to resuscitation, cardiac arrest, myocardial infarction, stroke, acute renal failure, acute liver failure, acute respiratory distress syndrome, sepsis or death from any case.
Thromboembolic events | up to five years
  Time from surgery to a thromboembolic event or death of any cause.
Minor outpatient complication | up to five years
  Time from discharge to minor outpatient complications, with death being considered as a competing risk event.
Length of hospital stay during index | an average of 10 days
  Days of hospitalization (from admission to last discharge with index case series)
Charges during index | an average of 10 days
  Sum of charges of all cases of the index case series

IPD SHARING:
Plan to Share IPD: No
The authors confirm that the data utilized in this study cannot be made available in the manuscript, the supplemental files, or in a public repository due to German data protection laws ('Bundesdatenschutzgesetz', BDSG). They are stored on a server of the BARMER Institute for Health System Research, to facilitate replication of the results. In general, access to data of statutory health insurance funds for research purposes is possible only under the conditions defined in German Social Law (SGB V § 287).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT06615999/Prot_SAP_000.pdf